CLINICAL TRIAL: NCT01047462
Title: Scandinavian Diverticulitis Trial. Laparoscopic Lavage vs Primary Resection as Treatment for Perforated Diverticulitis. A Randomized Prospective Multicenter Trial
Brief Title: Scandinavian Diverticulitis Trial
Acronym: SCANDIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Sykehuset Asker og Baerum (Other); Diakonhjemmet Hospital (Other); Sykehuset Ostfold (Other); Haukeland University Hospital (Other); Sykehuset Innlandet HF (Other); Karolinska University Hospital (Other); University Hospital, Linkoeping (Other); Helse Nord-Trøndelag HF (Other); Skane University Hospital (Other); Helse Nordmøre og Romsdal (Unknown); Ullevaal University Hospital (Other); Helse Stavanger HF (Other Government); Helse Nord (Industry); Uppsala University Hospital (Other); Centrallasarettet Västerås (Other); Sykehuset Buskerud HF (Other); Helsingborgs Hospital (Other); Vrinnevisjukhuset i Norrköping (Unknown); Eskilstuna Lasarettet (Other)
Responsible Party: Principal Investigator, Tom Oresland, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/177 (REK)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diverticulitis
MeSH Terms: conditions — Diverticulitis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic lavage (Active Comparator)
  Interventions: Procedure: Surgery for acute perforated diverticulitis
- Primary resection (Active Comparator)
  Interventions: Procedure: Surgery for acute perforated diverticulitis

INTERVENTIONS:
Procedure: Surgery for acute perforated diverticulitis — Primary resection vs laparoscopic lavage
  Other Names: Hartmann's procedure; Acute diverticulitis; Laparoscopic lavage; Primary resection

SUMMARY:
The purpose of this study is to determine whether laparoscopic lavage changes the rate of severe complications in patients with acute perforated diverticulitis who traditionally are treated with primary resection.

DETAILED DESCRIPTION:
Acute diverticulitis is a common disease in the western world. Perforation of the acute diverticulitis with peritonitis is a feared complication and standard treatment (primary sigmoid resection such as Hartmann's procedure) still has unsatisfactory results. Both mortality and morbidity are quite high. Several uncontrolled trials have reported a lower mortality and morbidity when acute perforated diverticulitis is treated with laparoscopic lavage instead of radical surgery. The investigators wish to conduct a randomized multicenter trial in Scandinavia in order to compare the rates of severe postoperative complications in acute perforated diverticulitis if treated by traditional primary sigmoid resection or by laparoscopic lavage. The investigators are planning to include all patients admitted to the participating hospitals with clinical and radiological findings of acute perforated diverticulitis.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* clinical suspicion of perforated diverticulitis with indication for urgent surgery
* CT scan with free air and findings suggesting diverticulitis
* patient tolerates general anaesthesia
* patients written consent

Exclusion Criteria:

* pregnancy
* bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-01 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
90 days complication rate | 90 days

SECONDARY OUTCOMES:
Quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tom Oresland, M.D., Ph.D., Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lorenskog, Norway

REFERENCES:
- [Derived] Azhar N, Johanssen A, Sundstrom T, Folkesson J, Wallon C, Korner H, Blecic L, Forsmo HM, Oresland T, Yaqub S, Buchwald P, Schultz JK; SCANDIV Study Group. Laparoscopic Lavage vs Primary Resection for Acute Perforated Diverticulitis: Long-term Outcomes From the Scandinavian Diverticulitis (SCANDIV) Randomized Clinical Trial. JAMA Surg. 2021 Feb 1;156(2):121-127. doi: 10.1001/jamasurg.2020.5618. PMID 33355658
- [Derived] Schultz JK, Wallon C, Blecic L, Forsmo HM, Folkesson J, Buchwald P, Korner H, Dahl FA, Oresland T, Yaqub S; SCANDIV Study Group. One-year results of the SCANDIV randomized clinical trial of laparoscopic lavage versus primary resection for acute perforated diverticulitis. Br J Surg. 2017 Sep;104(10):1382-1392. doi: 10.1002/bjs.10567. Epub 2017 Jun 20. PMID 28631827
- [Derived] Schultz JK, Yaqub S, Wallon C, Blecic L, Forsmo HM, Folkesson J, Buchwald P, Korner H, Dahl FA, Oresland T; SCANDIV Study Group. Laparoscopic Lavage vs Primary Resection for Acute Perforated Diverticulitis: The SCANDIV Randomized Clinical Trial. JAMA. 2015 Oct 6;314(13):1364-75. doi: 10.1001/jama.2015.12076. PMID 26441181